CLINICAL TRIAL: NCT04712474
Title: In-home Decluttering Augmentation of Group Cognitive-behavior Therapy for Hoarding Disorder: The Joining Forces Randomized Controlled Trial
Brief Title: In-home Decluttering Augmentation of Group CBT for HD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); City of Stockholm (Unknown); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Volen Ivanov, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-05798
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hoarding Disorder
Keywords: hoarding; clutter
MeSH Terms: conditions — Hoarding Disorder; Hoarding; Speech Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-home decluttering (Experimental): Study participants receive weekly sessions of in-home decluttering for 10 weeks.
  Interventions: Behavioral: In-home decluttering practice
- Delayed treatment (No Intervention): Study participants receive weekly session of in-home decluttering after a 10 week delay.

INTERVENTIONS:
Behavioral: In-home decluttering practice — The in-home decluttering intervention comprises 10, 1.5-hour home-visits over the course of 10 weeks.
  These home visits are personalized, goal-oriented and focused on decluttering. They include 1) a brief check-in, 2) guided unclutter time 3) a reflective period during which participants share their thoughts and objectives for the coming week, and 4) homework assignments.
  Arms: In-home decluttering

SUMMARY:
The primary aim of trial is to determine the clinical efficacy of in-home decluttering augmentation of group CBT for reducing hoarding severity in adults with HD. The trial takes place in Sweden.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) is the current evidence-based treatment for HD but the majority of sufferers remain symptomatic after CBT with impairing levels of clutter in their homes. Home visits, with a focus on in-home decluttering, have in previous research been shown to be a promising intervention when combined with CBT. However, augmenting CBT with subsequent home visits has not yet been tested in a randomized controlled trial (RCT). In response to this, in this trial, we aim to investigate the efficacy of a coordinated intervention, consisting of CBT and in-home decluttering for HD, in an RCT. In this trial, 90 participants with HD will initially receive 12 sessions of CBT through a psychiatric outpatient service. After CBT, participants will be randomized to receive either 10 home visits in 10 weeks, or to a wait list condition. Our hypothesis is that augmenting CBT with home visits will lead to a reduction in hoarding symptoms and clutter and improved daily functioning compared to wait list. We will also investigate the cost-economical aspects of the intervention. Results from this trial have the potential to reveal whether in-home decluttering should be added to CBT in order to reduce symptoms of hoarding and improve function in indviduals with HD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Hoarding disorder as primary psychiatric condition.
3. Willing and able to understand and complete consent and study procedures.
4. Living in the Stockholm county (Sweden) and within a 1-hour commute by public transport from the social services office.

Exclusion Criteria:

1. Concurrent CBT or having received CBT for HD during the last two years, for a minimum of 8 sessions including active strategies for reducing acquisition and practice of discarding with a qualified therapist or 8 previous in-home decluttering sessions with a qualified social worker.
2. Unable or unwilling to allow study staff into home for home assessment.
3. Animal hoarding or squalid (i.e. extremely unhygienic) home conditions that are deemed to put the personnel at risk during the in-home decluttering.
4. A diagnosis of organic brain disorder, intellectual disability, psychosis, bipolar disorder without stable medication or with symptoms within the last 6 months, anorexia nervosa or alcohol/substance dependence or abuse.
5. Major medical or neurological conditions that increase the risk of participation or that would prevent completing assigned behavioral practice tasks.
6. Immediate risk to self or others, requiring urgent medical attention, such as high suicidality risk.
7. Participant not able to read and communicate in Swedish.
8. Currently at high risk for eviction (for instance having received a "rättelseanmaning" by the housing company or Swedish court).
9. Potential participant lives in the same household as an already included participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Saving Inventory-Revised (SI-R) | Change from baseline (week 0) to post-treatment (week 10),
  The SI-R is a 23-item questionnaire with 3 sub-scales: 1) difficulty discarding, 2) excessive clutter, and 3) excessive acquisition.
Clutter Image Rating Scale (CIR) | Change from baseline (week 0) to post-treatment (week 10).
  Three sets of photographs, each comprising 9 photos of a room with varying levels of clutter. A selection is made as to which photograph best resembles the room of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Volen Ivanov, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst Stockholm, Huddinge, Sweden, 141 86, Stockholm, Sweden

REFERENCES:
- [Derived] Jagholm S, Lindstedt S, Andersson E, Mataix-Cols D, Fernandez de la Cruz L, Ruck C, Ivanov VZ. Study protocol for a randomized controlled trial of in-home decluttering augmentation of group cognitive-behavioral therapy for hoarding disorder: the Joining Forces Trial. Trials. 2023 Jul 29;24(1):483. doi: 10.1186/s13063-023-07509-4. PMID 37507772